CLINICAL TRIAL: NCT02072408
Title: Efficacy and Safety of Intravitreal Vascular Endothelial Growth Factor Trap-eye in Patients With Polyploidal Choroidal Vasculopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Kim's Eye Hospital (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-10-044-002
Record Dates: First submitted 2014-02-10; First posted 2014-02-26 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2014-02

CONDITIONS: Polypoidal Choroidal Vasculopathy Without Active Polyp
MeSH Terms: interventions — aflibercept

ARMS (1):
- polypoidal choroidal vasculopathy without polyp (Experimental)
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — 1. Three monthly intravitreal aflibercept (2mg) injections
  2. Five bimonthly intravitreal aflibercept (2mg) injections
  3. Rescue treatment: Verteporfin photodynamic therapy
     * Loss of five ETDRS letters or one Snellen line of vision from baseline
     * Presence of subretinal fluid or intraretinal fluid despite three consecutive (monthly or bimonthly) aflibercept injection
     * Presence of active polyp on indocyanine green angiography

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of aflibercept for treatment of polypoidal choroidal vasculopathy without active polyp.

ELIGIBILITY:
Inclusion Criteria:

* polypoidal choroidal vasculopathy without active polyp
* decreased visual acuity by subretinal fluid and hemorrhage involving foveal center

Exclusion Criteria:

* polypoidal choroidal vasculopathy with active polyp
* previous photodynamic therapy more than three times
* anti-VEGF injection within one month
* photodynamic therapy or intraocular steroid treatment within three months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-02; Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Change of best-corrected visual acuity (ETDRS letters) | 1 year

SECONDARY OUTCOMES:
presence of subretinal hemorrhage | during 1 year
  Total number of months when subretinal hemorrhage are detected on fundus photographs.
presence of fluid in macula evidenced by optical coherence tomography | during 1 year
  Total number of months when fluid in macula are detected on optical coherence tomography
change of indocyanine green angiography | during 1 year
  Change of indocyanine green angiography will include followings
  1. New appearance of polypoidal structure
  2. Any change in size of the greatest linear dimension of lesion
  3. Any change in size and activity of branching vascular network
Number of eyes which need rescue treatment (photodynamic therapy) | during 1 year
  In this study, photodynamic therapy will be performed as a rescue therapy according to the necessary criteria.
safety outcomes | one year
  frequency and severity of ocular adverse event

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam, Gyunggi-do
  - Konyang University Kim's Eye Hospital, Seoul
  - Samsung Medical Center, Seoul